CLINICAL TRIAL: NCT06292637
Title: Cognitive Behavioral and Faith Fellowship to Improve Thy Health (CB-FAITH) - A Feasibility and Acceptability Study
Brief Title: Cognitive Behavioral and Faith Fellowship to Improve Thy Health
Acronym: CB-FAITH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1484; 1R01HS029477-01 (AHRQ); A545000 (Other: UW Madison); NUR/FACULTY AFFAIRS/ADMIN (Other: UW Madison); Protocol Version 9/5/2025 (Other: UW Madison)
Record Dates: First submitted 2024-02-27; First posted 2024-03-05 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Depression
Keywords: faith-based intervention
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized stepped wedge design (R-SWD), a type of cluster randomized controlled trial, will be used to randomize a cluster (church groups with a group of 10 participants), not individual subjects.
  At the start of a R-SWD, all clusters begin as control groups. At certain time points during the course of the trial, some of the clusters are randomly selected to be switched to the CB-FAITH treatment, with all clusters eventually crossing over to receive the treatment. The sample will be comprised of 12 groups, each with 10 individuals (N=120).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- CB-FAITH treatment (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Faith Fellowship to Improve Thy Health (CB-FAITH)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Faith Fellowship to Improve Thy Health (CB-FAITH) — CB-FAITH is a behavioral depression intervention set inside a cognitive behavioral framework, and Afrocentric paradigm and informed by faith-based principles, designed to treat major depressive disorder among African American adults. The 13-treatment modules focus on increasing knowledge of depression and healthy coping behaviors. It is designed to be co-delivered by licensed mental health clinicians and pastors at churches.
  Arms: CB-FAITH treatment

SUMMARY:
Investigators will examine the efficacy of a faith-based depression intervention, in reducing symptoms of depression among African American adults in Wisconsin. Twelve church groups, each with 10 people (N=120) will be invited to participate. This intervention will be the first evidence-based, faith-based intervention designed for African Americans if validated.

DETAILED DESCRIPTION:
The randomized stepped wedge design (R-SWD) is a type of cluster randomized controlled trial in which the unit of randomization is a cluster (e.g., church groups with a group of 10 participants), not individual participants. At the start of a R-SWD, all clusters begin as control groups. At certain time points during the course of the trial, some of the clusters are randomly selected to be switched to the Cognitive Behavioral Faith Fellowship to Improve Thy Health (CB-FAITH) treatment, with all clusters eventually crossing over to receive the treatment.

Primary Aim 1: Examine efficacy of CB-FAITH in reducing symptoms of depression.

Secondary Aim 1: Examine moderating effects of religiosity on treatment effectiveness.

Secondary Aim 2: Evaluate satisfaction with CB-FAITH delivered in church settings.

Impact: CB-FAITH is poised to be the first evidence-based faith-based depression intervention designed for African American adults with depression. This community-prioritized research and transformative intervention has potential to reduce depression symptoms, reduce mental health disparities and advance health equity. Given the impact of COVID-19 pandemic, CB-FAITH is critically needed.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as an African American man or woman
* are ages 18 and older
* have symptoms of major depressive disorder, as evidenced by score of 10 and higher from the Patient Health Questionnaire-9 (PHQ-9).

Exclusion Criteria:

* major psychotic illnesses, such as schizophrenia;
* current participation in psychotherapy
* current suicidal ideations (trained staff will conduct a suicide risk assessment and facilitate referral for appropriate care).
* Medication stabilization. Eligible participants who report recent changes to their psychiatric medications (i.e., initiation of a new medication, change in dose or type of medication) will delay their study enrollment for a stabilization period of 4 weeks. Baseline data collection will be re-administered
* alcohol or drug dependence - those with alcohol or other drug dependence who have been clean and sober for 3 months will not be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire | baseline, weeks 6 and 12 during the intervention, and follow up at 3 and 6 months
  Patient Health Questionnaire-9 (PHQ-9) is a self-administered depression scale (5 minute completion time), which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day).
  Categories of depression symptoms are defined as none (score 0-4), mild (score 5-9), moderate (score 10-14), moderately severe (score 15-19), and severe (score ≥20). In addition to making criteria-based diagnoses of depressive disorders, the PHQ-9 is also a reliable and valid measure of depression severity.
Score on Quick Inventory of Depressive Symptomatology-clinician rated (QIDS-CR) | baseline, weeks 6 and 12 during the intervention, and follow up at 3 and 6 months
  The 16-item Quick Inventory of Depressive Symptomatology (QIDS) assesses depressive symptom severity and symptom change. Investigators will use the clinician rated QIDS-CR. Scores range from 0-27 and higher scores suggest higher severity of depression.

SECONDARY OUTCOMES:
Multidimensional Measure of Religious Involvement (MMRI) score | baseline, weeks 6 and 12 during the intervention, and follow up at 3 and 6 months
  Religiosity will be measured with the Multidimensional Measure of Religious Involvement (MMRI), a three-dimensional measure of religious involvement, consisting of organizational (frequency of service attendance), non-organizational (use of and frequency of nonorganized activities, such as watching religious programs on TV), and subjective religiosity (self-rated level of religiosity, such as significance of prayer and orientation toward God).
  It consists of 12 items and is self administered (5-10-minute completion time). Using Likert-scale responses, ranging from: 1 = very religious, 2 = fairly religious, 3 = not too religious, and 4 = not religious at all.
Client Satisfaction Inventory (CSI) score | approximately Week 13-16 (End of CB-FAITH classes)
  Client Satisfaction Inventory (CSI), an 8-item measure of satisfaction with counseling; total scores range from 8 to 32, with the higher number indicating greater satisfaction. The CSI will be self-administered.

CONTACTS AND LOCATIONS:
Overall Officials: Earlise Ward, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - University of Wisconsin - Madison, Madison, Wisconsin
  - Second Baptist Church, Madison, Wisconsin
  - The Board of Regents of the UW System, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No